CLINICAL TRIAL: NCT06149767
Title: Clinical Study of Adbelizumab Combined With Concurrent Chemoradiotherapy in Locally Advanced Cervical Cancer
Brief Title: Clinical Study of Adebrelimab Combined With Concurrent Chemoradiotherapy in Cervical Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-OBU-FJ-CA-001
Record Dates: First submitted 2023-09-14; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; adebrelimab
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adebrelimab Combined With Paclitaxel for Injection,cisplatin and radiotherapy (Experimental): Adebrelimab : 20 mg/kg, D1, intravenously, 30-60 min, Q3w. Paclitaxel for Injection: 150 mg/m2, D1 Cisplatin: 50 mg/m2, IV, D1, Q3w. Radiotherapy: pelvic dose: 6MV-X, 180cGy/ times 27 times; Brachydose: 192Ir, 700cGy/ time 4 times.
  Interventions: Drug: Adebrelimab

INTERVENTIONS:
Drug: Adebrelimab — The medication regimen for all enrolled patients is as follows, and the dose can be adjusted during treatment due to adverse reactions and other circumstances:
  Adebrelimab : 20 mg/kg, D1, intravenously, 30-60 min, Q3w. Paclitaxel for Injection: 150 mg/m2, D1 Cisplatin: 50 mg/m2, IV, D1, Q3w. Radiotherapy: pelvic dose: 6MV-X, 180cGy/ times 27 times; Brachydose: 192Ir, 700cGy/ time 4 times.
  First of all, after 2 cycles of concurrent chemoradiotherapy, the sequential chemotherapy combined with adbalizumab for 2-4 cycles, and the subsequent investigators selected Adbalizumab or other drugs to maintain the treatment according to the patient's situation or the patient's own will until the disease progressed or intolerable toxicity occurred or the subjects voluntarily withdrew from the study.adebrelimab until disease progression or intolerable toxicity or the subject voluntarily withdrew from the study。
  Other Names: Paclitaxel for Injection,cisplatin,radiotherapy

SUMMARY:
Prospective single-arm clinical study of adebrelimab combined with concurrent chemoradiotherapy in locally advanced cervical cancer

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of adebrelimab combined with concurrent chemoradiotherapy in locally advanced cervical cancer

ELIGIBILITY:
Inclusion Criteria:

1. The subjects understand and voluntarily participate in the study, sign the informed consent form (ICF), have good compliance, and cooperate with follow-up;
2. Female, 18 years of age ≤75 years of age on the date of signing the informed consent;
3. Cervical squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma confirmed by histopathology or cytology；
4. FIGO 2018 consists of patients with stage IIB - IVA. Note: Lymph nodes with confirmed metastasis are required for diagnosis of stage ⅢC1. Lymph node metastasis diagnosis can be confirmed by biopsy or imaging diagnosis, and the following criteria must be met for imaging diagnosis of lymph node metastasis: MRI or CT showing positive lymph nodes (minimum transverse diameter ≥15 mm)
5. Have not previously received any radical surgery, radiotherapy or systemic treatment (including investigational drugs) for cervical cancer, and have not received immunotherapy;
6. An American Eastern Oncology Collaboration (ECOG) score of 0 or 1 within 7 days prior to the first study intervention;
7. There is at least one measurable lesion that meets the requirements of RECIST v1.1 standard (tumor lesion with CT scan diameter ≥10mm, lymph node lesion with CT scan diameter ≥15mm, and scan layer thickness 5mm);
8. Expected survival ≥6 months;
9. The major organs function normally and meet the following criteria:

(1) Blood routine examination must meet:

1. Hemoglobin (Hb)≥90g/L
2. White blood cell count (WBC)≥3×109/L
3. Neutrophil count absolute value (ANC)≥1.5×109/L
4. Platelet count (PLT)≥100×109/L； (2) Biochemical examination shall meet the following standards:

a. Serum total bilirubin (TBIL) ≤1.5 × ULN (total bilirubin (BIL)≤3.0 mg/dL in patients diagnosed with Gilbert syndrome) b. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤3ULN c. Albumin (ALB) ≥3 g/dL d. Serum Cr≤1.5ULN, endogenous creatinine clearance ≥60ml/min (Cockcroft-Gault formula)； (3) The coagulation function test shall meet the following criteria:

1. International Standardized Ratio (INR) ≤1.5
2. Activated partial thromboplastin time (APTT) ≤1.5 ×ULN； 10. In potentially fertile women, serum or urine HCG negative for 72 hours prior to enlistment (postmenopausal women must be considered infertile for at least 12 months and a pregnancy test is not required for women who have been confirmed to have undergone tubal ligation), Female subjects of reproductive age and male subjects with a partner of a woman of reproductive age must consent to contraception for 24 weeks from the date of signing the informed consent to the last administration of the study drug.

Exclusion Criteria:

1. Subjects have histological subtypes other than those permitted by inclusion criteria 3;
2. Evidence of metastatic lesions according to RECIST 1.1 (including proximal L1 level or above or inguinal regional lymph nodes);
3. Have had a hysterectomy (defined as removal of the entire uterus) or had a hysterectomy as part of their initial treatment for cervical cancer;
4. Bilateral hydronephrosis, which the investigators judged could not be relieved by nephrostomy or ureteral stenting;
5. Patients with uncontrolled vaginal bleeding;
6. Previous allergy to any investigational drug ingredient;
7. Participate in clinical studies of other investigational drugs within 3 months prior to screening;
8. Other malignancies developed within 5 years prior to admission, excluding adequately treatable basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery;
9. Have any active autoimmune disease or history of autoimmune disease (such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitaritis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); Except for patients with vitiligo or childhood asthma/allergies that have healed and do not require any intervention as adults; Autoimmune mediated hypothyroidism treated with a steady dose of thyroid replacement hormone; Type 1 diabetes using steady doses of insulin;
10. A history of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation and allogeneic bone marrow transplantation;
11. Accompanied by serious heart, lung, liver, kidney disease; Having neurological or mental illness; Jaundice or digestive tract obstruction with severe infection;
12. Patients with hypertension who are not well controlled by antihypertensive drugs (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg); Or grade II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval ≥450ms for men and ≥470ms for women); According to NYHA criteria, patients with grade Ⅲ to Ⅳ cardiac insufficiency or left ventricular ejection fraction (LVEF) < 50% indicated by cardiac color ultrasound;
13. Urine routine suggests urinary protein ≥(++), or 24h urinary protein ≥1g or severe hepatic and renal insufficiency;
14. Patients with Crohn's disease and ulcerative colitis;
15. Subjects who have received systemic treatment with corticosteroids (>10 mg/ day of prednisone or other equivalent hormones) or other immunosuppressants within 2 weeks prior to initial dosing. In the absence of active autoimmune disease, inhaled or topical corticosteroids are permitted, as well as adrenal hormone replacement therapy at doses ≤10 mg/ day of prednisone efficacy;
16. Pregnant or lactating women, fertile subjects unwilling or unable to take effective contraceptive measures;
17. Those deemed unsuitable for inclusion by the researchers.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the 2-year PFS rate of adbelizumab combined with concurrent chemoradiotherapy in locally advanced cervical cancer. | up to 24 months
  To evaluate the 2-year PFS rate of adebrelimab combined with concurrent,Progression-free survival (PFS) as assessed by the investigators according to RECIST 1.1 criteria chemoradiotherapy in locally advanced cervical cancer
To evaluate the 2-year safety of adbelizumab combined with concurrent chemoradiotherapy in locally advanced cervical cancer. | up to 24 months
  evaluate the safety of adebrelimab combined with concurrent chemoradiotherapy in locally advanced cervical cancer,The security as assessed by the investigators according to CTCAE 5.0 criteria,All adverse events will also be rated based on the CTCAE version 5.0, and AEs greater than or equal to grade 3 will be statistically summarised.

SECONDARY OUTCOMES:
To evaluate the objective remission rate of adebrelimab combined with concurrent chemoradiotherapy in local advanced cervical cancer | up to 12 months
  To evaluate the objective remission rate of adebrelimab combined with concurrent chemoradiotherapy in local advanced cervical cancer
To evaluate the disease control rate of adebrelimab combined with concurrent chemoradiotherapy in local advanced cervical cancer | up to 24 months
  To evaluate the disease control rate of adebrelimab combined with concurrent chemoradiotherapy in local advanced cervical cancer
To evaluate the overall survival of adebrelimab combined with concurrent chemoradiotherapy in locally advanced cervical cancer | up to 24 months
  To evaluate the overall survival of adebrelimab combined with concurrent chemoradiotherapy in locally advanced cervical cancer

OTHER OUTCOMES:
A PD-L1 test | up to 12 months